CLINICAL TRIAL: NCT03661710
Title: Adherence to Prescribed Medication: Elucidating the Gap Between Guideline Recommendation and Real Life in Myocardial Infarction
Acronym: COMPLY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Andreas Kammerlander, PI, Medical University of Vienna
Other Study IDs: COMPLY-40400
Record Dates: First submitted 2018-09-01; First posted 2018-09-07 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Myocardial Infarction; Adherence, Medication
MeSH Terms: conditions — Myocardial Infarction; Medication Adherence | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Investigating Adherence to Standard of Care Medication and Cardiac Rehabilitation — Information from health care insurance providers on how many patients adhered to prescribed medication and how many underwent cardiac rehabilitation and how adherence influenced cardiovascular outcome will be retrieved

SUMMARY:
The aim of the study is to investigate the adherence to prescribed post-infarction medication and to cardiac rehabilitation in patients after acute myocardial infarction. In addition, their impact on cardiovascular events will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction
* Willingness to participate

Exclusion Criteria:

* Inclusion in an interventional study interfering with standard of care medication

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients after acute myocardial infarction requiring dual platelet inhibition
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Event | 3 years
  Composite of re-hospitalization due to acute MI, heart failure, stent thrombosis, fatal MI, and overall mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No